CLINICAL TRIAL: NCT02147639
Title: Effects of Sodium Nitrate on Blood Flow in Becker Muscular Dystrophy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NANO3
Record Dates: First submitted 2014-03-25; First posted 2014-05-28 (Estimated); Last update posted 2020-01-14 (Actual); Status verified 2014-05

CONDITIONS: Becker Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — sodium nitrate

ARMS (5):
- Sodium Nitrate (Experimental): Patients will ingest a single oral dose of sodium nitrate (~8.4 mmol)
  Interventions: Dietary Supplement: Sodium Nitrate
- Baseline (No Intervention): This is a baseline study visit, which will serve to assess inclusion and exclusion criteria, as well as provide untreated measurments of skeletal muscle blood flow and perfusion.
- Dose-escalation trial (Experimental): This is an optional study visit, where subjects will ingest twice the dose of sodium nitrate (~16.8 mmol).
  Interventions: Dietary Supplement: Sodium Nitrate - double dose
- Placebo-control trial (Placebo Comparator): This is an optional study visit, where patients will ingest a placebo.
  Interventions: Dietary Supplement: Placebo
- Increased exercise intensity (Experimental): This is an optional study visit, where patients will be asked to repeat all of the blood flow assessments, but the exercise intensity will be increased.
  Interventions: Procedure: Increased exercise intensity

INTERVENTIONS:
Dietary Supplement: Sodium Nitrate
  Arms: Sodium Nitrate
Dietary Supplement: Sodium Nitrate - double dose
  Arms: Dose-escalation trial
Dietary Supplement: Placebo
  Arms: Placebo-control trial
Procedure: Increased exercise intensity
  Arms: Increased exercise intensity

SUMMARY:
This study is intended to build on a growing body of literature showing a blood flow abnormality in patients with Becker muscular dystrophy. The investigators' laboratory recently showed that this blood flow abnormality could be corrected by a single oral dose of the drug Tadalafil (also known as Cialis). The investigators now wish to replicate these exciting results using a common nitric oxide donor (sodium nitrate).

DETAILED DESCRIPTION:
There are 2 phases to this research project: (1) an initial baseline study to confirm the blood flow abnormality in Becker muscular dystrophy, and (2) a subsequent brief treatment trial. There are also 3 optional study protocols: (A) dose-escalation trial, (B) placebo trial, and (C) increased exercise intensity trial.

The baseline study involves an intake history, physical examination, and phlebotomy for blood chemistries and DNA followed by non-invasive forearm blood flow studies (Near Infrared Spectroscopy, Doppler Ultrasound) before and after a brief bout of handgrip exercise (approximately 3-5 hours to complete). Blood flow studies will be performed with the subject's lower body enclosed in an airtight chamber. Blood flow and oxygen delivery to the forearm muscles will be measured before and during application of lower body negative pressure at rest and during handgrip exercise. Lower body negative pressure simulates the blood flow changes that normally occur when a person sits up after lying down.

The results of the baseline study will determine which patients meet preset eligibility criteria to participate in the medication phase of the study. These criteria include (1) normal kidney and liver function tests and normal BNP levels (the latter to exclude heart failure), and (2) abnormal blood flow responses to handgrip exercise.

Eligible patients will be asked to repeat the above laboratory procedures on a subsequent study day after receiving a single dose of sodium nitrate. Eligible patients will also be offered the option to repeat the above laboratory procedures on three subsequent study visits, where upon: (A) the dose of sodium nitrate is increased, (B) a placebo is ingested, and/or (C) the level of exercise in increased.

The investigators plan to enroll 20 adult men with Becker muscular dystrophy.

ELIGIBILITY:
Inclusion Criteria:

* Men 15-55 years of age with a pre-existing diagnosis of Becker Muscular Dystrophy by a clinical neurologist (based on clinical criteria plus previous muscle biopsy analysis and/or DNA analysis).

Exclusion Criteria:

* Any evidence of cardiopulmonary disease by history or by physical examination
* History of hypertension or blood pressure averaging ≥140/90 mmHg
* Diabetes mellitus or other systemic illness
* Heart failure by clinical exam, elevated BNP, or heart failure medication
* Serum creatinine ≥ 1.5 mg/dL
* Any history of substance abuse (including alcohol)
* Any history of psychiatric illness

Ages: 15 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Skeletal muscle blood flow | 24 hours after initial visit
  Skeletal muscle blood flow regulation will be assessed at each visit by near infrared spectroscopy and Doppler ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G Victor, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Heart Institute, Los Angeles, California, United States